CLINICAL TRIAL: NCT03395938
Title: Uncovering the Barriers of Colorectal Cancer Screening Amongst Siblings of Colorectal Cancer Patients Through a Randomised Control Trial.
Brief Title: Uncovering the Barriers of Colorectal Cancer Screening Amongst Siblings of Colorectal Cancer Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Health System, Singapore (Other)
Responsible Party: Principal Investigator, KER-KAN TAN, Consultant, Principal Investigator, National University Health System, Singapore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 2017/00172
Record Dates: First submitted 2017-05-14; First posted 2018-01-10 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Colorectal Cancer
Keywords: SCREENING
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Current practice (Placebo Comparator): "Intervention A" depicts current practices by having the research team educate the participants on the Ministry of Health Singapore screening guidelines akin to counselling sessions carried out during the patient's clinical consultation.
  Interventions: Behavioral: Current practice
- Proactive engagement (Active Comparator): "Intervention B" involves a series of proactive engagements in hope to spur patients into contacting their siblings and improve their receptiveness towards colorectal cancer screening.
  Interventions: Behavioral: Proactive engagement

INTERVENTIONS:
Behavioral: Proactive engagement — The engagements would include (1) a sealed envelope containing a cancer information sheet and an invitation letter directed towards siblings for them to contact the research team, (2) weekly phone reminders to the participants for a total of 4 weeks in a bid to remind participants of the need to convey the screening message to their siblings. The envelope will contain information on the various means for the siblings to contact the research team. These include communication means such as electronic mails (emails), telephone, hard copy returned mails through pre-paid envelopes, short messaging services (SMSs) or clinic consult.
  Arms: Proactive engagement
Behavioral: Current practice — This intervention depicts current practices by having the research team educate the participants on the Ministry of Health Singapore screening guidelines akin to counselling sessions carried out during the patient's clinical consultation. The research team would highlight that we would be happy to assist if necessary. The research team would then contact the patients in 4 weeks to check if they have communicated with their siblings and if they have gone for screening. We would also find out which method did they adopt to communicate with their siblings.
  Arms: Current practice

SUMMARY:
To determine amongst siblings of colorectal cancer patients:1. The knowledge, perception and barriers towards screening colonoscopy. 2. The current screening colonoscopy adoption rate. 3. If patients would engage them through active engagement by healthcare providers in a bid to improve their receptiveness towards and partake in colorectal cancer screening. 4. The method(s) that Colorectal cancer patients adopt to communicate with them. 5. If tailored interventions addressing logistical, psychological and cost barriers could increase the adoption of screening colonoscopy.

DETAILED DESCRIPTION:
Part I: Randomised control trial. Patients will be approached to participate in the study following recovery from their initial operation, after approximately three months, which often corresponds to the initial stages of adjuvant chemotherapy or active disease surveillance. Upon obtaining informed consent for the participant, the number of age appropriate siblings that are eligible for screening colonoscopy will be determined. Only siblings who have fulfilled the study inclusion criteria will be contacted. Siblings who accompany the participant for their follow-up appointment will directly be approached to participate in the qualitative component of the study. The Colorectal cancer patient will then be excluded from the Randomised control trial. However, given the findings of the preliminary study, most of the first degree relatives who came with the patients are the children and not siblings. As such the above mentioned scenario is unlikely. Participants will be enrolled into the randomised control trial and randomised to either "Intervention A" or "Intervention B". "Intervention A" depicts current practices by having the research team educate the participants on the Ministry of Health Singapore screening guidelines akin to counselling sessions carried out during the patient's clinical consultation. The research team would highlight that we would be happy to assist if necessary. The research team would then contact the patients in 4 weeks to check if they have communicated with their siblings and if they have gone for screening. The research team would also find out which method did they adopt to communicate with their siblings."Intervention B" involves a series of proactive engagements in hope to spur patients into contacting their siblings and improve their receptiveness towards colorectal cancer screening. The engagements would include (1) a sealed envelope containing a cancer information sheet and an invitation letter directed towards siblings for them to contact the research team, (2) weekly phone reminders to the participants for a total of 4 weeks in a bid to remind participants of the need to convey the screening message to their siblings. The envelope will contain information on the various means for the siblings to contact the research team. These include communication means such as electronic mails (emails), telephone, hard copy returned mails through pre-paid envelopes, short messaging services (SMSs) or clinic consult. A soft copy can also be given if requested by the patients.Once the participant has successfully contacted their siblings, the research team would inquire about the means of communication and the research team will proceed to invite the siblings to partake in the study. If the participant has yet contacted their siblings, the research team would inquire from participants as to why so. The research team will encourage the participant then to continue attempting to contact their siblings. Failing which at the end of 4 weeks, if the siblings remain not contactable, the participants will not be disturbed henceforth. Siblings who reject invitation to participate in the study will also not be contacted by the research team. Where possible, reasons for not being able to contact the siblings and rejections will be documented.

Siblings response rate will be determined in this study. The research team deem sibling replies as either "active" or "passive" by the way they use to contact the research team. "Active" approach would be for the siblings to contact the study team via the contact information provided to patients. "Passive" approach would be for the siblings to give verbal consent to the patient for the study team to contact them directly. This process is so tedious due to the Personal Data Protection Act (PDPA) that has been passed that prevent random calling of the siblings without informed consent.

ELIGIBILITY:
Inclusion Criteria for the siblings:

* Either Singaporean or Permanent Resident,
* Has a sibling who has been diagnosed with colorectal cancer
* Fulfilled the eligibility requirement to undergo screening colonoscopy as stipulated by Ministry of Health Singapore (At least aged 50 year or older or 10 years younger than when the index patient (below aged 60 year) was diagnosed with colorectal cancer)

Exclusion Criteria for the siblings include:

* Pre-existing family history of Familial Adenomatous Polyposis or Hereditary non-polyposis colorectal cancer
* Personal history of inflammatory bowel disease
* Personal history of colorectal cancer or colorectal polyps

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
The proportion of siblings that contacted the study team within 4 weeks from point of engagement by the index colorectal cancer patient. | 4 WEEKS
  The research team would like to compare the percentage response rates of siblings amongst the two intervention arms. A positive response would count as a sibling contacting the study team with their interest to undergo education by the research team on the topic of colorectal cancer screening.
  The research team would divide the method of positive response via
  1. "Active" approach would be for the siblings to contact the study team via the contact information provided to patients.
  2. "Passive" approach would be for the siblings to give verbal consent to the patient for the study team to contact them directly.

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No